CLINICAL TRIAL: NCT02699177
Title: In Vivo Measurements of Nasal Ciliary Beat Frequency by Using Interferometry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, SHOSEYOV DAVID, Dr., Hadassah Medical Organization
Other Study IDs: 0366-15-HMO-CTIL
Record Dates: First submitted 2015-12-29; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: ciliary beat frequency,
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — nasal brush biopsies, EM samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Suspected PCD but negative: CBF measurements:
  1. Patients with suspected PCD will have their nasal cavity photographed using a Sony-video camera that will record the reflected light of a green LED bulb.Ciliary beat frequency (CBF) will be calculated by interferometry using a program developed by the PI.
  2. Patients will undergo a nasal brush biopsies. The fresh biopsies will be analyzed by high-speed video microscopy to calculate CBF.
  3. The two methods will be compared.
  Interventions: Device: CBF measurements
- Suspected PCD but positive: CBF measurements:
  1. Patients with suspected PCD will have their nasal cavity photographed using a Sony-video camera that will record the reflected light of a green LED bulb.Ciliary beat frequency (CBF) will be calculated by interferometry using a program developed by the PI.
  2. Patients will undergo a nasal brush biopsies. The fresh biopsies will be analyzed by high-speed video microscopy to calculate CBF.
  3. The two methods will be compared.
  Interventions: Device: CBF measurements

INTERVENTIONS:
Device: CBF measurements — CBF measurements
  Other Names: Ciliary brush biopsy

SUMMARY:
1. Assessment of a high speed video camera with a green light source for the measurement of ciliary beat frequency (CBF) in the nasal airways of patients.
2. Assessments of the effect of drugs and other therapies on CBF using the study system.
3. Comparison of results with standard methods such as ciliary brush biopsies

DETAILED DESCRIPTION:
Background Mucociliary clearance of the airways depends on ciliary movement by ciliated cells that cover the entire airway and the sinuses. In many airway diseases the mucociliary clearance is affected by injury caused by smoke, viruses, other infectious organisms or genetic diseases that are called Primary Ciliary Dyskinesia (PCD).

The diagnosis of PCD is based on a combination of clinical findings such as bronchiectasis, chronic sinusitis, chronic otitis media and immotile sperms.

In addition, in tests performed in the pulmonary laboratory nasal nitric oxide levels may be low.

Samples obtained by nasal brush biopsy can be analyzed and the ciliary movement recorded by video microscopy. Ciliary beat frequency (CBF) can be calculated in freshly isolated samples but also after growing the tissue in cell culture.

Furthermore, ciliated cells can be analyzed by electron microscopy to detect defects in the microscopic structure of the cilia.

The major problem encountered by all these assays is that they are performed under in vitro conditions and not in the natural environment of the cells where the acidity (pH), temperature, electrolytes etc. may be very different.

Moreover, genetic testing is limited to mutations known to cause PCD, ruling out mutations not yet discovered.

Therefore a method is needed to unequivocally measure ciliary movement in the natural environment.

Goal

1. Assessment of a high speed video camera with a green light source for the measurement of ciliary beat frequency (CBF) in the nasal airways of patients.
2. Assessments of the effect of drugs and other therapies on CBF using the study system.

Methods The protocol has been approved by the local Institutional Review Board (IRB) of the Hadassah Medical Center, Jerusalem, Israel

Equipment:

1. High Speed High Video Microscope built to specifications needed for this study based on a commercially available high speed video system.
2. The green light source (LED) used consists of a spot of 3mm diameter and has an energy of 10 milli Watt ( equal to 1Kilowatt/square meter)
3. Video camera (manufactured by SONY Inc, Japan)

Patients:

Patients referred for ciliary brush biopsy will be asked to sign the informed consent and to be enrolled into the study.

Patients will be examined by having a high speed digital video camera placed close to the nasal cavity in order to photograph the area of interest. The camera lens will be off focus and the reflected light from the nasal mucosa will be recorded. This reflected light recording will be analyzed to obtain the CBF, heart rate and respiratory rate.

After the recording the patient will proceed to the nasal brush ciliary biopsy. The cells will be analyzed by a CBF will be calculated from several areas of the smear.

Safety measures:

All participating patients will wear a protective cover over their eyes during photography.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for Ciliary Brush Biopsy

Exclusion Criteria:

* Active nasal bleeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with suspected PCD
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Ciliary beat frequency (CBF) measured by high speed video microscopy | 5 minutes
  Ex vivo measurements of CBF analysing high speed video records of nasal brush biopsies
Ciliary beat frequency (CBF) measured by interferometry | 5 minutes
  In vivo measurements of CBF analysing the reflected light from the nasal cavity

CONTACTS AND LOCATIONS:
Overall Officials: David Shoseyov, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No